CLINICAL TRIAL: NCT02484898
Title: SEEQ™ Performance Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: SEEQ™ Performance Study
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2015-12

CONDITIONS: Arrhythmia Type Unknown

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SEEQ™ MCT/ECM System: SEEQ™ MCT/ECM monitoring for the detection of non-lethal cardiac arrhythmias.

SUMMARY:
The purpose of the Medtronic SEEQ™ Performance study is to build further evidence on the clinical and economic benefit of the Medtronic market-released SEEQ™ Mobile Cardiac Telemetry System/External Cardiac Monitor System (MCT/ECM).

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for a SEEQ™ MCT/ECM System for approved indications
* Patient is 18 years of age or older
* Patient is willing and able to provide consent and authorize the use and disclosure of health information
* Patient is willing and able to comply with the protocol

Exclusion Criteria:

* Patient has known allergy and/or hypersensitivity to adhesives or hydrogel.
* Patient has suspected potential life-threatening arrhythmias, or requires in-subject/in-hospital monitoring.
* Patient will undergo a medical procedure that would preclude full participate during the prescribed duration of the SEEQ™
* Patient has an implanted cardiac device, (e.g., pacemaker, Implantable Cardioverter Defibrillator, Cardiac Resynchronization Therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require monitoring for the detection of non-lethal cardiac arrhythmias such as, but not limited to, supraventricular tachycardias (for example, atrial fibrillation, atrial flutter, paroxysmal SVTs), ventricular ectopy, bradyarrhythmias, and conduction disorders.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SEEQ Performance Study Clinical Team, Study Director — Medtronic
Locations (9):
- United States (9):
  - Larkspur, California
  - Simi Valley, California
  - Aurora, Colorado
  - Clearwater, Florida
  - Palm Beach Gardens, Florida
  - Sebring, Florida
  - Rome, Georgia
  - Jackson, Mississippi
  - Henderson, Nevada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SEEQ™ MCT/ECM System
Started | 200
Completed | 182
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | SEEQ™ MCT/ECM System
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 91
Region of Enrollment [Number; unit: participants]
  United States | 200

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield of the SEEQ™ MCT/ECM System
Time Frame: 120 Days
Population: Subjects prescribed the SEEQ™ MCT/ECM monitoring for the detection of non-lethal cardiac arrhythmias
Measure: Number (95% Confidence Interval); unit: percentage of subjects with CRA
Arm/Group | SEEQ™ MCT/ECM System
Number analyzed (Participants) | 182
percentage of subjects with CRA | 85.7 [79.8 to 90.5]

ADVERSE EVENTS:
Arm/Group | SEEQ™ MCT/ECM System
Serious Adverse Events (participants affected / at risk) | 0/182
Other Adverse Events (participants affected / at risk) | 63/182
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEEQ™ MCT/ECM System (N=182)
Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin Irritation (Skin and subcutaneous tissue disorders) | 60 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less